CLINICAL TRIAL: NCT02123524
Title: A Phase III, Multi-centre, Randomized Trial to Compare Rivaroxaban With Placebo for the Treatment of Symptomatic Leg Superficial Vein Thrombosis
Brief Title: Rivaroxaban Anticoagulation for Superficial Vein Thrombosis
Acronym: RASET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCOG-2013-RASET
Record Dates: First submitted 2014-04-23; First posted 2014-04-25 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Symptomatic Superficial Vein Thrombosis
Keywords: Superficial Vein Thrombosis
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban 10mg tablet daily for 45 days
  Interventions: Drug: Rivaroxaban
- Control (Placebo Comparator): Placebo tablet daily for 45 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban
  Arms: Rivaroxaban
Drug: Placebo
  Arms: Control

SUMMARY:
This is a Phase III, randomized, placebo controlled, blinded, parallel two arm, multicentre trial that will compare rivaroxaban 10mg daily with placebo in patients with symptomatic leg Superficial Vein Thrombosis (> or = 5cm) that otherwise would not initially be treated with anticoagulant therapy.

DETAILED DESCRIPTION:
Patients with symptomatic superficial leg thrombosis will be randomized into two arms, a) rivaroxaban 10mg 1 tablet daily for 45 days or b) placebo to determine if rivaroxaban (10 mg once daily) is an effective and safe treatment for superficial vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

- Symptomatic Superficial Vein Thrombosis of the leg of ≥5 cm length (diagnosed clinically or with ultrasound)

Exclusion Criteria:

* Age <18 years
* Symptoms >42 days
* Receiving an anticoagulant for another indication (example: atrial fibrillation) when Superficial Vein Thrombosis started.
* Superficial Vein Thrombosis already treated with more than 3 days of anticoagulation (example. fondaparinux or Low Molecular Weight Heparin).
* Planned treatment of Superficial Vein Thrombosis with a course of anticoagulant therapy.
* Another indication for anticoagulant therapy (example. Deep Vein Thrombosis, Pulmonary Embolism, atrial fibrillation).
* Judged to require immediate ligation of the saphenofemoral junction or stripping of thrombosed varicose veins.
* proximal Deep Vein Thrombosis or Pulmonary Embolism within the past 12 months.
* Superficial Vein Thrombosis associated with sclerotherapy or an intravenous canula.
* A high risk of bleeding as evidenced by any of the following:

  1. Active bleeding
  2. Bleeding within the past 30 days due to a cause that has not fully resolved.
  3. Known or expected thrombocytopenia with a platelet count of less than 80,000 x 10 9/L.
  4. History of ever having had spontaneous intracranial bleeding, or any intracranial bleeding within the past 3 months.
  5. Receiving dual antiplatelet therapy (example. aspirin and clopidogrel).
* Elevated creatinine level is suspected and creatinine clearance has not been estimated, OR creatinine clearance (Cockcroft-Gault equation) of less than 30 ml/min.
* Clinically relevant hepatic disease (including Child-Pugh B and C) is known or suspected (example., associated with: International Normalized Ratio >1.7; total bilirubin >2 upper limit of normal; or Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) >3 times upper limit of normal).
* Ongoing requirement for systemic treatment with azole-antimycotics (except fluconazole), Human Immunodeficiency Virus (HIV) -protease inhibitors, or strong Cytochrome P450 3A4 (CYP3A4) inducers due to the potential interaction with rivaroxaban.
* Pregnant or lactating women, or at risk of becoming pregnant.
* Life expectancy less than 90 days
* Patient is unwilling or unable to comply with the protocol (example. unable to attend follow-up visits because of geographic inaccessibility).
* Participating in a competing clinical investigation and receiving any other investigational agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 90 days
  "Treatment failure" at 90 days (composite of: treated with non-study anticoagulant therapy; proximal Deep Vein Thrombosis or Pulmonary Embolism; surgery for Superficial Vein Thrombosis).
Safety | 90 Days
  Major bleeding within 90 days.

SECONDARY OUTCOMES:
Efficacy | Baseline,Day 7, Day 45 and Day 90
  The patient will self assess any change in leg pain using a Likert Scale.
Efficacy | Baseline and day 45
  Patients will rate any change in venous disease-specific quality of life (QOL) (VEINES-QOL and VEINES-Symptoms) and general health-related QOL (SF-36v2) at 45 days
Efficacy | Baseline, day 7, day 45 and day 90
  Any use of oral analgesics and oral/topical anti-inflammatory agents.
Safety | 90 days
  Death
Safety | 45 days
  major and minor bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MD, Principal Investigator — McMaster University/ Hamilton Health Sciences, Juravinski Hospital
Locations (11):
- Canada (11):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - St Josephs Healthcare, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - McMaster Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital Maisonneuve - Rosemount, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - St Mary's Hospital, Montreal, Quebec

REFERENCES:
- See also: Related Info — http://www.ocog.ca